CLINICAL TRIAL: NCT03568513
Title: Effect of Curcumin Food Supplement on Gut Microbiota in Children With Irritable Bowel Syndrome
Brief Title: Effect of Curcumin on Gut Microbiota in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Clinical & Translational Science Institute of Southeast Wisconsin (Other)
Responsible Party: Principal Investigator, Manu Sood, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1120142; UL1TR001436 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-06-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Curcumin; IBS and microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients in the treatment arm with weight between 35 kg to 50 kg will receive 50 mg capsule of curcumin twice a day (maximum dose 2.8 mg/kg/day, which is within the GRAS approved dose) and those over 50 kg in weight will receive three curcumin capsules a day (maximum dose 3 mg/kg/day, within GRAS recommended dose). Study duration will be 8 weeks.
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): Patients in the placebo arm will receive a capsule which has similar size, shape and color of the curcumin capsule. The placebo capsule will contain inert food powder. Study duration will be 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — The curcumin food supplement will be administered in the form of capsules. Participants in the treatment arm will take 50 mg twice or three times a day, depending on their body weight. Participants will take the curcumin capsules for eight weeks.
  Arms: Treatment
Dietary Supplement: Placebo — The placebo will be administered in the form of capsules. Participants in the placebo arm will take a capsule twice or three times a day, depending on their body weight. Participants will take the placebo capsules for eight weeks. The placebo capsule will be similar in size, shape and color to the curcumin capsule and they will contain inert food powder.
  Arms: Placebo

SUMMARY:
To evaluate the effect of curcumin food supplement on gut microbiota of children with irritable bowel syndrome (IBS) and to review any correlation between the changes in the microbiota with symptoms.

DETAILED DESCRIPTION:
This is a prospective, placebo-controlled, double blinded, randomized control trial. This study will evaluate the effect of curcumin food supplement on gut microbiota of children with irritable bowel syndrome. Curcumin is a commonly used spice in Asian cooking and has a very good safety profile. Developing preparation of this compound for targeted delivery in the GI tract would provide a novel way to treat common FGID. This study will provide preliminary data for future studies to evaluate the role of gut microbiota in the pathophysiology of pain predominant FGID and how food supplements can be used to manipulate the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 18 years old
* Fulfill the Rome IV criteria for diarrhea predominant IBS
* English speaking
* Able to swallow curcumin/placebo capsules

Exclusion Criteria:

* Weigh less than 35 kg
* On any form of dietary restrictions
* Taken probiotics one month before enrollment
* Antibiotic treatment one month before enrollment
* IBD
* Celiac disease
* Peptic ulcer disease
* H. Pylori gastritis
* Abnormality of gastrointestinal tract
* Previous abnormal endoscope
* Previous abdominal surgeries
* Gall stones
* Biliary tract obstructions
* Liver pathologies
* Liver failure
* Active GI infection
* Positive stool cultures
* Drug or alcohol abuse
* Concomitant immunological/hematological/neoplastic/heart/ renal/pulmonary condition
* Any other medical condition or taking any form of drug(s) which can explain the current symptoms
* Take oral or intravenous drugs which could have potential drug interaction with curcumin
* Lactating or pregnant or planning to become pregnant
* Developmental delay
* Parents that are developmentally delayed
* Have a diet high in curcumin/turmeric

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Alteration in Gut Microbiota | 8 weeks
  To study the alteration in gut microbiota with 8-week curcumin dietary supplementation in children with IBS between the ages of 10 yrs to 18 yrs

SECONDARY OUTCOMES:
Comparison of GI Symptoms | 8 weeks
  To compare the GI symptoms at baseline and after 8-weeks of curcumin dietary supplementation we will be using a previously validated Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) questionnaire (Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther 1997; 11(2): 395-402). This questionnaire measures symptom severity and includes a scale of "none" to "very severe" or "very happy to very unhappy" or "not at all" to "completely" as well as "often/occasionally/never." The maximum achievable score is 500 and mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300 and >300 respectively. Higher scores means worse outcome and vice versa. At the end of the 8-weeks curcumin supplementation any absolute or relative decrease in the total score in comparison to baseline will considered as improvement in outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Manu Sood, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03568513/ICF_001.pdf